CLINICAL TRIAL: NCT00673920
Title: A Randomized, Double-Blind, Parallel-Group, International Study to Evaluate the Safety and Efficacy of Ocrelizumab Given As a Single Infusion or Dual Infusion Compared With Placebo in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate Therapy
Brief Title: A Study to Evaluate Ocrelizumab Compared With Placebo in Patients With Rheumatoid Arthritis Who Have an Inadequate Response to Methotrexate Therapy
Acronym: FEATURE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on analysis of results and consideration of available treatments, the overall benefit to risk profile of ocrelizumab was not favorable in RA.
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT4394g; WA20496
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- Placebo (Placebo Comparator): Participants received matching placebo:
  * on Day 15 of Cycle 1 (Participants who were administered OCR 400 mg on Day 1 of a Cycle 1 in combination with Methotrexate)
  * on both Days 1 and Day 15 of Cycle 1 (Participants who were randomized to the Placebo + Methotrexate group)
  Interventions: Drug: Methotrexate; Drug: Placebo
- Ocrelizumab 400mg (Experimental): Participants received Ocrelizumab 400mg in combination with Methotrexate on Day 1, Cycle 1.
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab
- Ocrelizumab 200mg (Experimental): Participants received Ocrelizumab 200 mg in combination with Methotrexate on Day 1 and Day 15, Cycle 1.
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab
- Ocrelizumab 200mg/ Ocrelizumab 200mg (Experimental): Participants who received two 200 mg infusions of Ocrelizumab + Methotraxate during Cycle 1 were re-randomized (1:1 randomization ratio) to receive two infusions of 200 mg Ocrelizumab + Methotraxate during Cycle 2
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab
- Ocrelizumab 200mg/ Ocrelizumab 400mg (Experimental): Participants who received two 200 mg infusions of Ocrelizumab + Methotraxate during Cycle 1 were re-randomized (1:1 randomization ratio) to receive a single infusion of 400 mg Ocrelizumab + Methotraxate during Cycle 2
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab
- Ocrelizumab 400mg/ Ocrelizumab 400mg (Experimental): Participants who received single 400mg infusions of Ocrelizumab + Methotraxate during Cycle 1 received a infusion of 400 mg Ocrelizumab + Methotraxate during Cycle 2
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab
- Placebo/ Ocrelizumab 200mg (Experimental): Participants who received placebo during Cycle 1 were re-randomized (1:1 randomization ratio) to receive two infusions of 200 mg Ocrelizumab + Methotraxate during Cycle 2
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab; Drug: Placebo
- Placebo/ Ocrelizumab 400mg (Experimental): Participants who received placebo during Cycle 1 were re-randomized (1:1 randomization ratio) to receive single infusion of 400 mg Ocrelizumab + Methotraxate during Cycle 2
  Interventions: Drug: Methotrexate; Drug: Ocrelizumab; Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Oral or parenteral repeating dose
Drug: Ocrelizumab — Ocrelizumab was administered as a slow intravenous (iv) infusion during each course as either 200 mg on Day 1 and Day 15 (OCR 200×2) or as 400 mg given on Day 1 (OCR 400×1).
  Ocrelizumab was administered in combination with Methotrexate.
  Arms: Ocrelizumab 200mg; Ocrelizumab 200mg/ Ocrelizumab 200mg; Ocrelizumab 200mg/ Ocrelizumab 400mg; Ocrelizumab 400mg; Ocrelizumab 400mg/ Ocrelizumab 400mg; Placebo/ Ocrelizumab 200mg; Placebo/ Ocrelizumab 400mg
Drug: Placebo — Intravenous repeating dose
  Arms: Placebo; Placebo/ Ocrelizumab 200mg; Placebo/ Ocrelizumab 400mg

SUMMARY:
This study will evaluate the efficacy and safety of ocrelizumab, compared to placebo, in patients with active rheumatoid arthritis who have an inadequate response to methotrexate therapy. Patients will be randomized 2:2:1 to receive 1) infusions of ocrelizumab 200mg iv on Days 1 and 15, 2) infusions of ocrelizumab 400mg iv on Day 1 and placebo iv on Day 15, or 3) infusions of placebo iv on Days 1 and 15. At the end of the placebo-controlled treatment period at 24 weeks, patients in groups 1 and 3 will be re-randomized to receive either a single infusion of 400mg iv ocrelizumab or 2 infusions of 200mg iv ocrelizumab, and group 2 will receive a second single infusion of 400mg iv ocrelizumab. All patients will receive a stable dose of concomitant methotrexate (7.5-25mg/week) throughout the study. The anticipated time on study treatment is 1-2 years. Target number of patients to be enrolled in this trial is 300.

ELIGIBILITY:
Inclusion criteria:

* Adult patients, ≥ 18 years of age
* Active rheumatoid arthritis
* Inadequate treatment with any DMARD other than methotrexate

Exclusion criteria:

* Rheumatic autoimmune disease or inflammatory joint disease other than rheumatoid arthritis
* Concurrent treatment with any DMARD other than methotrexate
* Previous treatment with any cell-depleting therapies
* Any surgical procedure in past 12 weeks, or planned within 48 weeks after baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2008-04-24 (Actual); Primary Completion 2009-10-26 (Actual); Study Completion 2009-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dummer, M.D., Study Director — Genentech, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Emery P, Rigby W, Tak PP, Dorner T, Olech E, Martin C, Millar L, Travers H, Fisheleva E. Safety with ocrelizumab in rheumatoid arthritis: results from the ocrelizumab phase III program. PLoS One. 2014 Feb 3;9(2):e87379. doi: 10.1371/journal.pone.0087379. eCollection 2014. PMID 24498318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening was completed within 28 days prior to randomization. This may have been extended by an additional 56 days, up to a maximum of 84 days, if washout from the respective disease modifying anti-rheumatic drugs (DMARDs) or if immunization was required.
Period: Baseline up to Week 48
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Started | 64 | 117 | 133 | 0 | 0 | 0 | 0 | 0
Completed | 60 | 114 | 126 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Refused treatment | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Insufficient therapeutic response | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Violation of selection criteria at entry | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Administrative/Other | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event/intercurrent illness | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Period: Week 24 to Week 48
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Started | 0 | 0 | 0 | 61 | 61 | 109 | 29 | 28
Completed | 0 | 0 | 0 | 60 | 61 | 106 | 28 | 28
Not Completed | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0
Not completed — Adverse event/intercurrent illness | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Failure to return | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Insufficient therapeutic response | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adminstrative/Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics not provided for Participants who were re-randomized at Week 24 (Cycle 2)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg | Total
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0 | 312
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (11.45) | 52.3 (11.14) | 53.0 (11.15) |  |  |  |  |  | 52.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 93 | 105 |  |  |  |  |  | 254
  Male | 8 | 24 | 26 |  |  |  |  |  | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 22 | 24 |  |  |  |  |  | 56
  Not Hispanic or Latino | 54 | 95 | 107 |  |  |  |  |  | 256
  Unknown or Not Reported | 0 | 0 | 0 |  |  |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 2 |  |  |  |  |  | 8
  Asian | 4 | 13 | 10 |  |  |  |  |  | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  |  |  |  | 0
  Black or African American | 9 | 9 | 9 |  |  |  |  |  | 27
  White | 44 | 85 | 99 |  |  |  |  |  | 228
  More than one race | 0 | 0 | 0 |  |  |  |  |  | 0
  Unknown or Not Reported | 4 | 7 | 11 |  |  |  |  |  | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Response
Description: ACR20 response: greater than or equal to (≥) 20% improvement in tender or swollen joint counts and 20% improvement in 3 of the following 5 criteria: 1) Physician's global assessment of disease activity, 2) participant assessment of disease activity, 3) Patient Assessment of Pain (visual analog scale [VAS]), 4) participant assessment of functional disability via a Health Assessment Questionnaire (HAQ), and 5) erythrocyte sedimentation rate (ESR) at each visit.
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Ocrelizumab 200mg - Cycle 1: Participants received Ocrelizumab 200 mg in combination with Methotrexate on Day 1 and Day 15, Cycle 1.
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 28.1 [17.1 to 39.1] | 37.6 [28.8 to 46.4] | 52.7 [44.1 to 61.2] |  |  |  |  |

2. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score 28 (DAS28) Remission (DAS28 < 2.6)
Description: The DAS28 was derived from assessments of erythrocyte sedimentation rate (ESR) measured in millimeters per hour (mm/h), tender joint count on 28 joints (TJC28), swollen joint count on 28 joints (SJC28), and Patient's Global Assessment of disease activity according to 100--millimeter (mm) Visual Analog Scale (VAS). DAS28 score was calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. DAS28 score could range from 0 to 10, where higher score represented higher disease activity. The change from Week 24 to Week 40 was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 3.1 | 4.3 | 5.3 |  |  |  |  |

3. Secondary Outcome: Change in DAS28 From Baseline
Description: The DAS28 was derived from assessments of erythrocyte sedimentation rate (ESR) measured in millimeters per hour (mm/h), tender joint count on 28 joints (TJC28), swollen joint count on 28 joints (SJC28), and Patient's Global Assessment of disease activity according to 100--millimeter (mm) Visual Analog Scale (VAS). DAS28 score was calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. DAS28 score could range from 0 to 10, where higher score represented higher disease activity. The change from Week 24 to Week 40 was averaged among all participants, where negative changes indicated an improvement in disease activity. The change is the difference in adjusted mean change from baseline in DAS28 between ocrelizumab 400 x 1 and ocrelizumab 200 x 2 with placebo.
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 49 | 104 | 119 | 0 | 0 | 0 | 0 | 0
Units on scale | -0.79 (1.293) | -1.60 (1.374) | -1.67 (1.320) |  |  |  |  |

4. Secondary Outcome: European League Against Rheumatism (EULAR) Response Rates (Categorical DAS Responders)
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Percentage of Participants
  Week 4 No Response | 62.5 | 62.4 | 58.0 |  |  |  |  |
  Week 4 Moderate Response | 37.5 | 33.3 | 38.9 |  |  |  |  |
  Week 4 Good Response | 0 | 4.3 | 3.1 |  |  |  |  |
  Week 8 No Response | 70.3 | 52.1 | 48.1 |  |  |  |  |
  Week 8 Moderate Response | 28.1 | 39.3 | 42.0 |  |  |  |  |
  Week 8 Good Response | 1.6 | 8.5 | 9.9 |  |  |  |  |
  Week 12 No Response | 68.8 | 41.9 | 35.9 |  |  |  |  |
  Week 12 Moderate Response | 29.7 | 49.6 | 54.2 |  |  |  |  |
  Week 12 Good Response | 1.6 | 11.1 | 9.9 |  |  |  |  |
  Week 16 No Response | 68.8 | 39.3 | 35.1 |  |  |  |  |
  Week 16 Moderate Response | 29.7 | 49.6 | 47.3 |  |  |  |  |
  Week 16 Good Response | 1.6 | 11.1 | 17.6 |  |  |  |  |
  Week 20 No Response | 68.8 | 41.0 | 30.5 |  |  |  |  |
  Week 20 Moderate Response | 26.6 | 48.7 | 51.1 |  |  |  |  |
  Week 20 Good Response | 4.7 | 10.3 | 18.3 |  |  |  |  |
  Week 24 No Response | 73.4 | 44.4 | 38.9 |  |  |  |  |
  Week 24 Moderate Response | 21.9 | 41.0 | 47.3 |  |  |  |  |
  Week 24 Good Response | 4.7 | 14.5 | 13.7 |  |  |  |  |

5. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response
Description: The ACR50 response at any time was defined as >/=50% improvement compared to baseline in TJC (assessed on 68 joints) and SJC (assessed on 66 joints); and 50% improvement compared to baseline in 3 of the following 5 criteria, respectively: 1) Patient's global assessment of disease activity according to 100-mm VAS, 2) Physician's global assessment of disease activity according to 100-mm VAS, 3) participant's global assessment of pain according to 100-mm VAS, 4) Participant's assessment of functional ability via HAQ-DI, and 5) Acute phase reactant (ESR in mm/h or CRP in mg/dL).
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 7.8 | 18.8 | 30.5 |  |  |  |  |

6. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response
Description: The ACR70 response at any time was defined as >/=70% improvement compared to baseline in TJC (assessed on 68 joints) and SJC (assessed on 66 joints); and 70% improvement compared to baseline in 3 of the following 5 criteria, respectively: 1) Patient's global assessment of disease activity according to 100-mm VAS, 2) Physician's global assessment of disease activity according to 100-mm VAS, 3) participant's global assessment of pain according to 100-mm VAS, 4) Participant's assessment of functional ability via HAQ-DI, and 5) Acute phase reactant (ESR in mm/h or CRP in mg/dL).
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 1.6 | 6.8 | 7.6 |  |  |  |  |

7. Secondary Outcome: Change From Baseline in the Individual Parameters of the ACR Core Set
Description: Change in the scores of the following parameters of ACR core set relative to respective baseline scores was measured: SJC (28 and 66 joints) and TJC (28 and 66 joints), patient's global assessment and physician's global assessment based on disease activity (both are expressed by VAS [0 = no disease activity to 100 = maximum disease activity]), HAQ (based on HAQ disability index [HAQDI]) which included 8 domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities) rated on a 4-point scale (0=without any difficulty to 3=unable to do), where the sum of scores was divided by the number of domains with a score for a total possible score of 0 (best) to 3 (worst), pain assessment using a VAS ranging from score 0 (no pain) to 100 (unbearable pain).
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number; unit: Units on a scale
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Units on a scale
  SJC | -4.6 | -7.5 | -8.7 |  |  |  |  |
  TJC | -8.2 | -10.2 | -12.0 |  |  |  |  |
  Patient's global assessment | -7.6 | -21.2 | -24.3 |  |  |  |  |
  Physician's global assessment | -16.0 | -24.3 | -26.0 |  |  |  |  |
  Patient's pain assessment | -8.0 | -17.2 | -21.0 |  |  |  |  |
  HAQ-DI | -0.2 | -0.4 | -0.5 |  |  |  |  |

8. Secondary Outcome: Change From Baseline in the Individual Parameters of the ACR Core Set: C-Reactive Protein (CRP) Concentration
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number; unit: mg/dL
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
mg/dL | -0.2 | -1.0 | -0.8 |  |  |  |  |

9. Secondary Outcome: Change From Baseline in the Individual Parameters of the ACR Core Set: Erythrocyte Sedimentation Rate (ESR)
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number; unit: mm/hr
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
mm/hr | -3.0 | -14.2 | -11.1 |  |  |  |  |

10. Secondary Outcome: Percentage of Participants With a Reduction of Greater Than or Equal to 0.25 Units in the HAQ-DI Score
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 37.5 [25.6 to 49.4] | 55.6 [46.6 to 64.6] | 58.8 [50.3 to 67.2] |  |  |  |  |

11. Secondary Outcome: Change in SF-36 Subscale and Summary Scores From Baseline
Description: Improved, change > 5.42; Unchanged, -5.42 <= Change <= 5.42; Worsened, change < -5.42
Time Frame: Week 24
Population: ITT Population (original randomization)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Percentage of Participants
  Mental Component Summary Category Improved | 42.0 | 34.9 | 36.6 |  |  |  |  |
  Mental Component Summary Category Unchanged | 38.0 | 50.0 | 51.2 |  |  |  |  |
  Mental Component Summary Category Worsened | 20.0 | 15.1 | 12.2 |  |  |  |  |
  Physical Component Improved | 44.0 | 45.3 | 53.7 |  |  |  |  |
  Physical Component Unchanged | 42.0 | 51.9 | 42.3 |  |  |  |  |
  Physical Component Worsened | 14.0 | 2.8 | 4.1 |  |  |  |  |

12. Secondary Outcome: Change in FACIT-F Fatigue Assessment From Baseline
Description: The FACIT-Fatigue score was calculated according to a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participants fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). Clinically relevant improvement is defined as a greater than or equal to (≥)5-point change from Baseline.
Time Frame: Baseline, Weeks 4, 12, and 24
Population: ITT Population (original randomization)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 64 | 117 | 131 | 0 | 0 | 0 | 0 | 0
Units on a scale
  Baseline: number analyzed (Participants) | 63 | 117 | 130 | 0 | 0 | 0 | 0 | 0
  Baseline | 25.13 (10.616) | 25.33 (11.313) | 24.74 (11.161) |  |  |  |  |
  Week 4: number analyzed (Participants) | 63 | 117 | 131 | 0 | 0 | 0 | 0 | 0
  Week 4 | 28.94 (11.371) | 28.60 (11.231) | 30.71 (11.136) |  |  |  |  |
  Week 12: number analyzed (Participants) | 55 | 114 | 128 | 0 | 0 | 0 | 0 | 0
  Week 12 | 28.42 (12.015) | 32.09 (12.368) | 33.09 (10.903) |  |  |  |  |
  Week 24: number analyzed (Participants) | 50 | 108 | 127 | 0 | 0 | 0 | 0 | 0
  Week 24 | 28.47 (12.406) | 31.38 (11.346) | 33.18 (11.011) |  |  |  |  |

13. Secondary Outcome: Percentage of Participants Achieving an ACR20 Response
Description: as for outcome 1
Time Frame: Week 48
Population: Study extension period included all participants who were re-randomized at Week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 0 | 0 | 0 | 61 | 61 | 109 | 29 | 28
Percentage of Participants |  |  |  | 59.0 | 54.1 | 56.9 | 44.8 | 42.9

14. Secondary Outcome: Percentage of Participants Achieving an ACR50 Response
Description: as for outcome 5
Time Frame: Week 48
Population: Study extension period included all participants who were re-randomized at Week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 0 | 0 | 0 | 61 | 61 | 109 | 29 | 28
Percentage of Participants |  |  |  | 36.1 | 27.9 | 34.9 | 20.7 | 14.3

15. Secondary Outcome: Percentage of Participants Achieving an ACR70 Response
Description: as for outcome 6
Time Frame: Week 48
Population: Study extension period included all participants who were re-randomized at Week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 0 | 0 | 0 | 61 | 61 | 109 | 29 | 28
Percentage of Participants |  |  |  | 19.7 | 16.4 | 19.3 | 6.9 | 7.1

16. Secondary Outcome: Percentage of Participants Achieving DAS28 Remission (DAS28 < 2.6)
Time Frame: Week 48
Population: Study extension period included all participants who were re-randomized at Week 24.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
Number analyzed (Participants) | 0 | 0 | 0 | 61 | 61 | 109 | 29 | 28
Percentage of Participants |  |  |  | 13.1 | 3.3 | 11.0 | 6.9 | 3.6

17. Secondary Outcome: Cmax: Maximum Observed Serum Concentration of Ocrelizumab Following First Infusion
Time Frame: Week 24, 48
Population: Placebo population was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Ocrelizumab 200mg - Cycle 2: Participants who received two 200 mg infusions of Ocrelizumab + Methotraxate in Cycle 2
- Ocrelizumab 400mg - Cycle 1: Participants received Ocrelizumab 400mg in combination with Methotrexate on Day 1, Cycle 1.
- Ocrelizumab 400mg - Cycle 2: Participants who received a single infusion of 400 mg Ocrelizumab + Methotraxate in Cycle 2
Arm/Group | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg - Cycle 2 | Ocrelizumab 400mg - Cycle 1 | Ocrelizumab 400mg - Cycle 2
Number analyzed (Participants) | 120 | 85 | 107 | 183
μg/mL | 73.1 (63.8) | 67.7 (27.0) | 133 (38.5) | 137 (45.4)

18. Secondary Outcome: Csecond: Maximum Observed Serum Concentration of Ocrelizumab Following Second Infusion
Time Frame: Day 15 of Cycles 1 and 2
Population: Population included all participants who received second Ocrelizumab infusion.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ocrelizumab 200mg - Cycle 1 | Ocrelizumab 200mg - Cycle 2
Number analyzed (Participants) | 117 | 83
μg/mL | 71.7 (18.0) | 77.6 (27.4)

ADVERSE EVENTS:
Time Frame: From baseline up to 17 months
Description: Re-randomized Safety Population: All patients (including those not re-randomized at Week 24) who received any part of the second course and provided at least one assessment of safety prior to Week 48 were included in the Re-randomized Safety Population.
Arm/Group | Placebo | Ocrelizumab 400mg | Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 200mg | Ocrelizumab 200mg/ Ocrelizumab 400mg | Ocrelizumab 400mg/ Ocrelizumab 400mg | Placebo/ Ocrelizumab 200mg | Placebo/ Ocrelizumab 400mg
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/117 | 0/131 | 0/61 | 0/61 | 1/109 | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 5/64 | 3/117 | 2/131 | 5/61 | 5/61 | 10/109 | 3/29 | 0/28
Other Adverse Events (participants affected / at risk) | 32/64 | 59/117 | 80/131 | 46/61 | 49/61 | 86/109 | 20/29 | 22/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Ocrelizumab 400mg (N=117) | Ocrelizumab 200mg (N=131) | Ocrelizumab 200mg/ Ocrelizumab 200mg (N=61) | Ocrelizumab 200mg/ Ocrelizumab 400mg (N=61) | Ocrelizumab 400mg/ Ocrelizumab 400mg (N=109) | Placebo/ Ocrelizumab 200mg (N=29) | Placebo/ Ocrelizumab 400mg (N=28)
BRONCHIECTASIS (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 5 (5) | 5 (5) | 9 (9) | 3 (3) | 0 (0)
MYCOBACTERIUM ABSCESSUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Ocrelizumab 400mg (N=117) | Ocrelizumab 200mg (N=131) | Ocrelizumab 200mg/ Ocrelizumab 200mg (N=61) | Ocrelizumab 200mg/ Ocrelizumab 400mg (N=61) | Ocrelizumab 400mg/ Ocrelizumab 400mg (N=109) | Placebo/ Ocrelizumab 200mg (N=29) | Placebo/ Ocrelizumab 400mg (N=28)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 12 (12) | 16 (16) | 5 (5) | 14 (14) | 14 (14) | 2 (2) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5) | 3 (3) | 7 (7) | 6 (6) | 1 (1) | 4 (4) | 3 (3) | 2 (2)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 7 (7) | 7 (7) | 1 (1) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
INFUSION RELATED REACTION (General disorders) | 7 (7) | 25 (25) | 28 (28) | 19 (19) | 17 (17) | 28 (28) | 5 (5) | 6 (6)
FATIGUE (General disorders) | 4 (4) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 4 (4) | 10 (10) | 6 (6) | 2 (2) | 6 (6) | 1 (1) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 6 (6) | 3 (3) | 3 (3) | 2 (2) | 7 (7) | 3 (3) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
HEADACHE (Nervous system disorders) | 4 (4) | 5 (5) | 7 (7) | 5 (5) | 5 (5) | 6 (6) | 2 (2) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 7 (7) | 4 (4) | 5 (5) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.